CLINICAL TRIAL: NCT03425110
Title: The Modified Ketogenic Diet for the Treatment of Pharmacoresistant Epilepsy in Adults: an Observational Cohort Study
Brief Title: The Modified Ketogenic Diet for the Treatment of Pharmacoresistant Epilepsy in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Birmingham and Solihull Mental Health NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 173471
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Modified Ketogenic Diet

SUMMARY:
The Modified Ketogenic Diet for the Treatment of Pharmacoresistant Epilepsy in Adults: an Observational Cohort Study

DETAILED DESCRIPTION:
Epilepsy is a common neurological condition. Unfortunately, just over 30% of patients with epilepsy (PWE) do not become seizure free with anti-epileptic drugs. Some patients may be suitable for epilepsy surgery. Alternative established treatments include vagal nerve stimulation and the ketogenic diet in children. The evidence base for the use of ketogenic diet in adults is limited. There are a few prospective studies and no randomised control trial to date.

This study is a prospective observational cohort study for adult patients with drug resistant epilepsy who are not suitable for resective epilepsy surgery. The intervention is a modified ketogenic diet. The carbohydrate load will be between 20-30gm per day. Blood ketones and blood sugars will be monitored. The primary outcome measure is seizure frequency at 12 months. There are a number of secondary outcome measures including tolerability, seizure severity, quality of life, lipid profiles and health care utilisation.

ELIGIBILITY:
The study will have no formal inclusion/exclusion criteria as it is purely observational and it will be the clinical team's decision as to whether or not people are seen by the dietary clinic based on established dietary clinic protocols.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult outpatients with pharmacoresistant epilepsy referred to and accepted by the epilepsy clinic will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-07-21 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
50% responder rate | Twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Manny Bagary, Dr, Study Director — Consultant Epileptologist and Neuropsychiatrist
Locations (1):
- Complex Epilepsy Service, The Barberry, BSMHFT, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No